CLINICAL TRIAL: NCT01972737
Title: A Phase I Study of Guanylyl Cyclase C (GCC)-Encoding Replication-Deficient Human Type 5 Recombinant Adenovirus Vaccine (Ad5-hGCC-PADRE) in Stage I and II Colon Cancer Patients
Brief Title: Phase I Study of Ad5-hGCC (Human Guanylyl Cyclase C)-PADRE in Stage I/II Colon Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sidney Kimmel Cancer Center at Thomas Jefferson University (Other)
Responsible Party: Sponsor
Organization: Thomas Jefferson University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 13S.462; SAP #4100051723 (Other Grant/Funding Number: Pennsylvania Department of Health); JT 2657 (Other: JeffTrial Number)
Record Dates: First submitted 2013-10-24; First posted 2013-10-30 (Estimated); Last update posted 2025-05-02 (Actual); Status verified 2025-05

CONDITIONS: Colon Cancer
Keywords: Vaccine; Colon cancer; safety; tolerability; antibody responses; T cell responses
MeSH Terms: conditions — Colonic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Ad5-hGCC-PADRE Vaccine (Experimental): Active vaccine
  Interventions: Biological: Ad5-hGCC-PADRE vaccine

INTERVENTIONS:
Biological: Ad5-hGCC-PADRE vaccine — A single intramuscular dose (100 billion virus particles) of Ad5-hGCC-PADRE vaccine.

SUMMARY:
The purpose of this study is to determine the safety, tolerability and ability to stimulate hGCC-specific antibody and killer T cell immune responses of an Ad5-hGCC-PADRE vaccine in stage I and stage II Caucasian and African American colon cancer patients.

DETAILED DESCRIPTION:
There is an unmet need for improved therapeutic paradigms in colorectal cancer, the 3rd leading cause of cancer and 2nd leading cause of cancer mortality worldwide. This need is underscored by the populations in jeopardy, including the ~100 million people in the US over 50 y that have a 1:8 risk associated with a disease-specific mortality of 50%. Mortality reflects metastatic disease: ~50% of patients initially present with regional or distant metastases, while ~20% present with occult metastases. Beyond the general population risk, there is an established stage-specific difference in outcomes in pN0 (node negative) African Americans with colorectal cancer, who exhibit ~40% excess mortality attributable to race. Reductions in mortality have been hampered by the absence of effective chemo-, radio-, and immuno- therapeutic approaches to metastatic disease. In that context, immunotherapy has been disappointing, in part, reflecting the absence of antigens that are tumor-specific, immunogenic, and universally associated with neoplasia. Moreover, the gap in survival between African Americans and Caucasians specifically reflects the inability to identify those with occult metastases who are at increased risk for developing recurrent disease.

This study advances an emerging paradigm in colorectal cancer cell detection and eradication, employing GCC as a molecular marker and immunological target. GCC is a protein whose expression is normally restricted to intestinal epithelial cells, but universally expressed by metastatic colorectal tumors. We have clinically validated the detection of occult metastases in lymph nodes by quantifying GCC mRNA (messenger RNA) by reverse transcriptase (RT)-PCR (qRT-PCR). This study revealed that occult metastases were the most powerful independent predictors of survival in pN0 patients. Further, there is a disproportionate burden of occult disease in African American, compared to Caucasian, patients. This new molecular staging platform provides a unique opportunity to identify occult metastases underlying racial disparities in disease recurrence, which could be prevented by tumor-targeted immunotherapy.

In the absence of ideal tumor antigens, immunotherapy has been directed to tissue-specific proteins. Barriers to employing self-antigens include tolerance, which limits anti-tumor immunity, and autoimmunity. The present study advances an emerging paradigm exploiting immunological compartmentalization of mucosally-restricted antigens to generate systemic antitumor immunity without autoimmunity. Asymmetry in immunological cross-talk between compartments, wherein systemic T and B cell responses rarely extend to mucosae, suggest that proteins normally expressed in mucosae, but which are expressed systemically by tumors, may serve as vaccine targets for metastases. Advantages of these cancer mucosa antigens include unique systemic immunoreactivity profiles supporting highly effective durable antitumor immunity in the context of absent immunological cross-talk between compartments restricting autoimmunity. Here, this paradigm will be advanced employing the tumor marker GCC, which induces immune responses that oppose metastatic colorectal cancer in preclinical models, without autoimmunity. This study will define the safety and immunological efficacy of adenoviral GCC vaccine in African American and Caucasian pN0 colon cancer patients with excess recurrence risk reflecting occult lymph node metastases identified by GCC qRT-PCR. This study will be the first step in translating GCC into a vaccine for the secondary prevention of metastases in African American and Caucasian colorectal cancer patients.

ELIGIBILITY:
Inclusion Criteria:

* Male and Female African American or Caucasian subjects older than 18 years of age. Race will be defined by the subject.
* Stage I or stage II (pN0) colon cancer within 3 years of surgery
* Competent immune system, defined by the ability to make a delayed type hypersensitivity (DTH) reaction to at least one of the following: candida, mumps, tetanus or trichophyton
* Adequate renal, liver, and bone marrow functions:

Serum creatinine ≤ 2.0 mg/dl, Hemoglobin ≥ 10.0 g/dl WBC (white blood cells) ≥ 3,000 /mm3, platelet count ≥ 100,000/mm3, total bilirubin ≤2.0 mg/ml, and albumin ≥ 3.0 g/dl

* Lymph node specimens available for quantification of occult metastases
* Minimum of 2 months and maximum of 36 months since surgery
* No clinical or laboratory evidence of local or systemic recurrence at entry to the study
* Expected survival of at least 6 months
* Karnofsky performance status ≥ 80 (ECOG 0 or 1)
* Willingness and ability to understand and give informed consent and follow the procedures described in the protocol

Exclusion Criteria:

* Failure to meet any of the inclusion criteria above
* Rectal cancer
* Prior chemotherapy/radiotherapy/immunotherapy/experimental medications for colon cancer
* Prior splenectomy
* Concurrent use of systemic steroids or immunosuppressive drugs (Note: topical or inhaled aerosol steroid therapies are not contraindicated for participation in the study)
* HIV-positive by ELISA, confirmed by Western blot
* Active autoimmune diseases that the Investigator considers would interfere with an immunologic response (e.g., systemic lupus erythematosus, multiple sclerosis or ankylosing spondylitis)
* Other malignancy within 5 years except curatively treated non-melanomatous skin cancer and curatively treated carcinoma in situ of the uterine cervix, or early stage (stage A or B1) prostate cancer
* Medically-proven inflammatory bowel disease
* Has at the time of enrollment, serious infection or other serious medical condition that implies a survival of less than six months
* Pregnancy or lactation (serum B-human chorionic gonadotropin test must be negative in fertile women at screening visit). Subjects will be asked to use contraception during conduct of the study.
* Past medical history of serious reaction to adenovirus vaccine
* Mental handicap
* Chronic diarrhea >6 times per day

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2013-10; Primary Completion 2014-06-03 (Actual); Study Completion 2016-01-13 (Actual)

PRIMARY OUTCOMES:
Adverse events | Continuous for 6 months after vaccination.
  Quantify treatment-emergent and related acute and sub-acute adverse events, serious adverse events, and Grade 3 and 4 non-laboratory abnormalities for safety assessments during the 6-month period after the injection of Ad5-hGCC-PADRE.
Antibody responses | One month following vaccination.
  Determine whether Ad5-hGCC-PADRE induces an antibody response to GCC at 1 month following vaccination with Ad5-hGCC-PADRE.

SECONDARY OUTCOMES:
T cell responses | One month following vaccination.
  Determine whether Ad5-hGCC-PADRE induces a T cell response to GCC at 1 month following vaccination.
Persistent immunological responses | Three and six months after vaccination.
  Determine whether Ad5-hGCC-PADRE induces antibody and/or T cell responses to GCC that persist at 3 months and 6 months following vaccination.

OTHER OUTCOMES:
Occult metastases and immune responses | One, three, and six months following vaccination.
  Determine whether antibody and/or T cell responses to GCC following vaccination with Ad5-hGCC-PADRE are related to occult metastases in regional lymph nodes quantified by GCC qRT-PCR.
Race and immune responses | One, three and six months following vaccination.
  Determine whether antibody and/or T cell responses to GCC following vaccination with Ad5-hGCC-PADRE are related to race.
Time to recurrence and disease-free survival and immune responses | Annually for 5 years from the time of vaccination
  Determine whether antibody and/or T cell responses to GCC following vaccination with Ad5-hGCC-PADRE are related to time to recurrence and/or disease-free survival during the 5-year period after the injection of Ad5-hGCC-PADRE.

CONTACTS AND LOCATIONS:
Overall Officials: Scott A Waldman, MD, PhD, Study Director — Thomas Jefferson University
Locations (1):
- Thomas Jefferson University, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Background] Waldman SA, Hyslop T, Schulz S, Barkun A, Nielsen K, Haaf J, Bonaccorso C, Li Y, Weinberg DS. Association of GUCY2C expression in lymph nodes with time to recurrence and disease-free survival in pN0 colorectal cancer. JAMA. 2009 Feb 18;301(7):745-52. doi: 10.1001/jama.2009.141. PMID 19224751
- [Background] Snook AE, Magee MS, Marszalowicz GP, Schulz S, Waldman SA. Epitope-targeted cytotoxic T cells mediate lineage-specific antitumor efficacy induced by the cancer mucosa antigen GUCY2C. Cancer Immunol Immunother. 2012 May;61(5):713-23. doi: 10.1007/s00262-011-1133-0. Epub 2011 Nov 6. PMID 22057677
- [Background] Snook AE, Li P, Stafford BJ, Faul EJ, Huang L, Birbe RC, Bombonati A, Schulz S, Schnell MJ, Eisenlohr LC, Waldman SA. Lineage-specific T-cell responses to cancer mucosa antigen oppose systemic metastases without mucosal inflammatory disease. Cancer Res. 2009 Apr 15;69(8):3537-44. doi: 10.1158/0008-5472.CAN-08-3386. Epub 2009 Apr 7. PMID 19351847
- [Background] Snook AE, Huang L, Schulz S, Eisenlohr LC, Waldman SA. Cytokine adjuvanation of therapeutic anti-tumor immunity targeted to cancer mucosa antigens. Clin Transl Sci. 2008 Dec;1(3):263-4. doi: 10.1111/j.1752-8062.2008.00054.x. PMID 19956776
- [Background] Snook AE, Stafford BJ, Eisenlohr LC, Rothstein JL, Waldman SA. Mucosally restricted antigens as novel immunological targets for antitumor therapy. Biomark Med. 2007 Jun;1(1):187-202. doi: 10.2217/17520363.1.1.187. PMID 20477468
- [Background] Snook AE, Stafford BJ, Li P, Tan G, Huang L, Birbe R, Schulz S, Schnell MJ, Thakur M, Rothstein JL, Eisenlohr LC, Waldman SA. Guanylyl cyclase C-induced immunotherapeutic responses opposing tumor metastases without autoimmunity. J Natl Cancer Inst. 2008 Jul 2;100(13):950-61. doi: 10.1093/jnci/djn178. Epub 2008 Jun 24. PMID 18577748
- [Derived] Snook AE, Baybutt TR, Xiang B, Abraham TS, Flickinger JC Jr, Hyslop T, Zhan T, Kraft WK, Sato T, Waldman SA. Split tolerance permits safe Ad5-GUCY2C-PADRE vaccine-induced T-cell responses in colon cancer patients. J Immunother Cancer. 2019 Apr 23;7(1):104. doi: 10.1186/s40425-019-0576-2. PMID 31010434
- [Derived] Myers RE, Wolf T, Shwae P, Hegarty S, Peiper SC, Waldman SA. A survey of physician receptivity to molecular diagnostic testing and readiness to act on results for early-stage colon cancer patients. BMC Cancer. 2016 Oct 3;16(1):766. doi: 10.1186/s12885-016-2812-1. PMID 27716119